CLINICAL TRIAL: NCT02256462
Title: Pediatric Crohn's Disease AdalImumab Level-based Optimization Treatment (PAILOT) Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Schneider Children's Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Amit Assa, Dr, Schneider Children's Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAILOT
Record Dates: First submitted 2014-09-26; First posted 2014-10-03 (Estimated); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interventional (Experimental): Adalimumab levels and antibodies will be obtained with every laboratory examination (every 2 months, except for the first 2 visits). Dose or interval adjustment will be performed as followed:when trough levels results taken prior to ADA injection are above 5 µg/ml no change in dosing is required. Detectable levels below 5 µg/ml will result in interval decrease to every week. If levels are still below 5 µg/ml dose will be increased to 40 mg (in patients receiving less than 40 mg). Undetectable levels below 0.3µg/ml will be followed by antibodies (ATAs) measurement. If ATAs are persistently above 8 µg/ml the patient will discontinue the study. If ATAs are below 8 µg/ml ADA intervals will be decreased to every week.
  Interventions: Drug: Adalimumab
- Clinical (No Intervention): Adalimumab levels and antibodies will be requested based on physician judgment when there are signs of loss of response (LOR). Dose and interval adjustment will be performed according to clinical measures: Following physician decision trough levels and ATAs will be collected and further adjustment may be considered according to results. Interval adjustment will be performed as described for the interventional arm.
  LOR is defined as PCDAI equal or higher than 10 or CRP higher than 0.5 mg/dl (5mg/l) and/or Fecal calprotectin higher than 150 mcg/gr (If lower than 150 at randomization).

INTERVENTIONS:
Drug: Adalimumab — Eligible patients are those who are planned to start Adalimumab (ADA). Patients will be randomized at the first screening visits to either group 1 (interventional) or group 2 (clinical). Eligible patients, will start induction treatment (weeks 0,2) with ADA (> 40kg 160/80/40 mg every 2 weeks or < 40 kg 100/50/25 mg for m2 body surface area every 2 weeks). Interventions will start from the 4th injection for responding patients only (based on levels taken prior to the third injection). Responding patients will continue to the maintenance phase in which they will receive ADA every 2 weeks, either 40 mg or 25 mg/m2. At screening, and every 2 months all patients will be examined and have height, weight, PCDAI performed as well as comprehensive laboratory examinations.
  Other Names: Humira
  Arms: Interventional

SUMMARY:
Objectives: To examine the effect of drug level-based personalized treatment of adalimumab in children with Crohn's disease. Design: A prospective, randomized, open label study. Setting: Pediatric gastroenterology centers. Participants: Children 6 year to 17 years who are diagnosed with CD and are planned to receive adalimumab treatment. Main outcome measures: Pediatric Crohn's Activity Index (PCDAI) at 48 and 72 weeks. Secondary outcome measures: Corticosteroids free remission rates and on adalimumab at 48 and 72 weeks. The effect of routine adalimumab drug monitoring-based treatment on trough levels and anti-adalimumab antibodies during therapy.

DETAILED DESCRIPTION:
The efficacy of adalimumab in inducing and maintaining remission in both adults and children with moderate-to-severe Crohn's Disease has been demonstrated in multiple clinical trials. Despite efforts to optimize treatment, approximately 40% of patients who initially respond to anti-TNF ultimately lose response. Measurement of adalimumab (ADA) drug levels and antibodies to adalimumab (ATAs) in patients has been shown to assist decision making in patients who have lost response during the course of treatment. This approach is based on the observations showing that higher ADA concentrations are associated with higher treatment efficacy and that loss of response is primarily attributed to either undetectable drug levels or to the presence of high titers of ATAs. Existing data is mostly based on retrospective cohort studies, nevertheless, the concept of routine therapeutic drug monitoring in-order to improve efficacy is still evolving. Recently, preliminary results of the Trough level Adapted infliXImab Treatment (TAXIT) study, performed in adult IBD patients, have failed to demonstrate superiority of level-based treatment over clinically-based treatment regarding rates of response over time. Nevertheless, it is premature to conclude that patients do not benefit from a tailored approach as the reported abstract did not stratify patients according to type of disease (CD vs. ulcerative colitis) and as some significant advantages such as reduced rate of antibodies and reduction of CRP were described in the level-based arm. Anti-TNF treatment in pediatric patients may differ from adults due to a higher risk for developing the rare hepatosplenic T cell lymphomas (HSCTL) in young males treated with combination therapy including thiopurines and anti-TNF agents. Concomitant therapy (using immunomodulators, mainly azathioprine) which has demonstrated superiority over mono-therapy has become a standard of care in moderate to severe CD in adults. In-view of the concerns of pediatric gastroenterologist from concomitant therapy-induced adverse events the option to improve efficacy of mono-therapy by guiding it according to drug monitoring is further appealing. Therefore, our aim is to assess the efficacy of routine therapeutic drug monitoring based treatment in pediatric CD patients in a prospective randomized control trial. We hope that this study will further contribute to the understanding of the potential benefits of therapeutic drug monitoring based management in pediatric patients treated with anti-TNF agents.Hypothesis:

We hypothesize that by routine measuring of ADA trough levels and ATAs titers we will achieve higher and stable trough levels resulting in greater corticosteroid free remission rates and decreased LOR rates. We assume that this will be associated with lower frequencies of ATAs. We further assume that the intervention will reduce the need for alteration of treatment schemes by adding immunomodulators or by switching treatment within class or out of class.

Objectives:

This is ADA therapy optimization study in patients starting or receiving ADA due to active disease.

1. Primary Efficacy Objective: To evaluate the effect of routine ADA drug monitoring-based treatment, in comparison to clinically-based monitoring on disease activity.
2. Secondary Objective: To evaluate the effect of routine ADA drug monitoring-based treatment on trough levels and ATAs during therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Crohn's disease
2. Age 6-17 (inclusive)
3. Naïve to biologics
4. Informed consent
5. Neg. TB-Test, negative HBV- S Ag
6. Negative stool culture, parasites and clostridium toxin

Inclusion criteria Comments:

1. Patients receiving corticosteroids may be included if on taper-down scheduled to be completed by week 10.
2. Partial enteral nutrition, accounting for less than 50% of daily required calories, may be supplied as needed.
3. Patients receiving antibiotics must cease use of antibiotics within the 14 days of receiving the first injection. Excluding immunomodulators (azathioprine/6MP and methotrexate), any other targeted therapy for crohn's disease (i.e 5-ASA) must be stopped prior to ADA first injection. Immunomodulators will be required to be stopped either prior to first ADA injection or at 6 months following ADA initiation.

Exclusion Criteria:

1. Pregnancy.
2. Renal Failure.
3. Current abscess or perforation of the bowel.
4. Small bowel obstruction within the last 6 months.
5. Fixed non inflammatory stricture with related symptoms.
6. Complicated or heavily draining perianal fistula (indolent non draining or minimally draining fistula are not an exclusion criteria).
7. Prior treatment with infliximab or adalimumab.
8. Previous malignancy.
9. Sepsis or active bacterial infection.
10. Surgery related to Crohn's disease in the previous 8 weeks.
11. Positive Hepatitis B surface antigen or evidence for TB.
12. IBD unclassified.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Loss of response (LOR) during treatment. | Week 72
  Patients with loss of response are defined as those with a good initial clinical response to anti-TNFα, with a later clinical and biochemical relapse defined as PCDAI≥10 (for patients in remission) or an increase of 15 points PCDAI from post induction baseline and CRP> 0.5mg/dl and/or calprotectin>150µgr/gr

SECONDARY OUTCOMES:
Corticosteroids free complete clinical remission, on ADA, | 48 and 72 weeks
  Patients with PCDAI<10, and quiescent disease by physician global assessment (PGA).
Trough levels | 8, 16, 32, 48, 72 weeks
  Mean adalimumab trough levels
Antibodies to adalimumab | 8, 16, 32, 48, 72 weeks
  Presence of antibodies to adalimumab (ATAs)
Anthropometric indices | 0, 4, 8, 16, 24, 32, 40, 48, 56, 64, 72, weeks
  Anthropometric indices (weight, height, BMI) and growth assessment during scheduled visits
Laboratory markers | 0, 4, 8, 16, 24, 32, 40, 48, 56, 64, 72, weeks
  Laboratory surrogate markers (CBC, ESR, CRP, albumin, fecal calprotectin) during scheduled visits
Adverse events | 4, 8, 16, 24, 32, 40, 48, 56, 64, 72, weeks
  Medication associated adverse events
The need for treatment modification during therapy | Week 72
  Addition of immunomodulator, switch within/out of class
Disease activity defined by PCDAI | 48 and 72 weeks
  Pediatric Crohn's Disease Activity Index

CONTACTS AND LOCATIONS:
Overall Officials: Raanan Shamir, MD, Study Chair — Tel Aviv University
Locations (1):
- Schneider Children's Hospital, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hanauer SB, Sandborn WJ, Rutgeerts P, Fedorak RN, Lukas M, MacIntosh D, Panaccione R, Wolf D, Pollack P. Human anti-tumor necrosis factor monoclonal antibody (adalimumab) in Crohn's disease: the CLASSIC-I trial. Gastroenterology. 2006 Feb;130(2):323-33; quiz 591. doi: 10.1053/j.gastro.2005.11.030. PMID 16472588
- [Background] Colombel JF, Sandborn WJ, Rutgeerts P, Enns R, Hanauer SB, Panaccione R, Schreiber S, Byczkowski D, Li J, Kent JD, Pollack PF. Adalimumab for maintenance of clinical response and remission in patients with Crohn's disease: the CHARM trial. Gastroenterology. 2007 Jan;132(1):52-65. doi: 10.1053/j.gastro.2006.11.041. Epub 2006 Nov 29. PMID 17241859
- [Background] Karmiris K, Paintaud G, Noman M, Magdelaine-Beuzelin C, Ferrante M, Degenne D, Claes K, Coopman T, Van Schuerbeek N, Van Assche G, Vermeire S, Rutgeerts P. Influence of trough serum levels and immunogenicity on long-term outcome of adalimumab therapy in Crohn's disease. Gastroenterology. 2009 Nov;137(5):1628-40. doi: 10.1053/j.gastro.2009.07.062. Epub 2009 Aug 5. PMID 19664627
- [Background] Paul S, Moreau AC, Del Tedesco E, Rinaudo M, Phelip JM, Genin C, Peyrin-Biroulet L, Roblin X. Pharmacokinetics of adalimumab in inflammatory bowel diseases: a systematic review and meta-analysis. Inflamm Bowel Dis. 2014 Jul;20(7):1288-95. doi: 10.1097/MIB.0000000000000037. PMID 24831559
- [Derived] Matar M, Shamir R, Lev-Zion R, Broide E, Weiss B, Ledder O, Guz-Mark A, Rinawi F, Cohen S, Topf-Olivestone C, Shaoul R, Yerushalmi B, Assa A. The Effect of Adalimumab Treatment on Linear Growth in Children With Crohn Disease: A Post-hoc Analysis of the PAILOT Randomized Control Trial. J Pediatr Gastroenterol Nutr. 2020 Aug;71(2):237-242. doi: 10.1097/MPG.0000000000002728. PMID 32324651
- [Derived] Matar M, Shamir R, Turner D, Broide E, Weiss B, Ledder O, Guz-Mark A, Rinawi F, Cohen S, Topf-Olivestone C, Shaoul R, Yerushalmi B, Ben-Horin S, Assa A. Combination Therapy of Adalimumab With an Immunomodulator Is Not More Effective Than Adalimumab Monotherapy in Children With Crohn's Disease: A Post Hoc Analysis of the PAILOT Randomized Controlled Trial. Inflamm Bowel Dis. 2020 Oct 23;26(11):1627-1635. doi: 10.1093/ibd/izz294. PMID 31793630
- [Derived] Assa A, Matar M, Turner D, Broide E, Weiss B, Ledder O, Guz-Mark A, Rinawi F, Cohen S, Topf-Olivestone C, Shaoul R, Yerushalmi B, Shamir R. Proactive Monitoring of Adalimumab Trough Concentration Associated With Increased Clinical Remission in Children With Crohn's Disease Compared With Reactive Monitoring. Gastroenterology. 2019 Oct;157(4):985-996.e2. doi: 10.1053/j.gastro.2019.06.003. Epub 2019 Jun 10. PMID 31194979